CLINICAL TRIAL: NCT00001917
Title: M2 Receptor Measurements in Aging and in Alzheimer's Disease
Brief Title: Brain Imaging in Elderly People and Individuals With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990073; 99-M-0073
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Alzheimer's Disease; Healthy
Keywords: Positron Emission Tomography; Physostigmine; Visual Stimulation; Cholinergic Stimulation; [F-18] FP-TZIP; Aging; Alzheimer's Disease; Visual Activation
MeSH Terms: conditions — Alzheimer Disease | interventions — FP-TZTP

INTERVENTIONS:
Drug: O15
Drug: [F-18] FP-TZTP

SUMMARY:
The purpose of this study is to use brain imaging technology to study the effects of aging and Alzheimer's Disease (AD) on a specific type of brain receptor.

The brain is made up of cells called neurons. The neurons communicate with one another and secrete chemicals called neurotransmitters. The neurotransmitters bind to specific sites on other neurons called receptors. Acetylcholine (ACh) is a neurotransmitter that binds to ACh receptors. In both aging and AD, the number of neurons that secrete ACh decreases and the function of some ACh receptors changes. This study will use positron emission tomography (PET) scans of the brain to study the effects of age and AD on muscarinic type 2 [M2], a type of ACh receptor.

Participants in this study will be injected with a radioactive tracer (ligand [F-18] FP-TZTP) which binds to [M2] receptors. Participants will then undergo a PET scan in order for the density and function of [M2] receptors to be studied.

DETAILED DESCRIPTION:
The Geriatric Psychiatry Branch (GPB) of the National Institute of Mental Health (NIMH) proposes to study the effect of aging and Alzheimer's Disease (AD) on muscarinic type 2 (M2) receptor density and function using the ligand [F-18] FP-TZTP. M2 receptors are primarily autoreceptors found on acetylcholine (ACh) neurons, and are lost along with ACh neurons in aging and AD, particularly in the cerebral cortex. As we near completion of the study of the young versus the old, we would like to add a few more healthy subjects to achieve better gender balance, continue the accrual of Alzheimer's patients and expand the Protocol to include its natural scientific progression. Quantification of M2 receptors with a single FP-TZTP scan as we are currently performing with 99-M-0073 provides a measure of the number of cholinergic receptors in the brain, but not their capacity to release acetylcholine into the synapse. To test this capacity requires a second TZTP scan and the use of an agent that alters acetylcholine concentrations in the synapse. Non-human primate studies performed here (1) have found PET scans with FP-TZTP to be sensitive to changes in acetylcholine synapse concentrations, as a result of competition, in response to the adminstration of the acetylinesterase inhibitor physostigmine. We would like to use physostigmine in all groups; young, older normal, and Alzheimer's patients to infer differences in capacity to release acetylcholine.

ELIGIBILITY:
INCLUSION CRITERIA:

Healthy males and females between 20-100 years old and volunteers with AD.

AD volunteers must meet the NINCDS-ADRDA criteria for possible, probable, or definite AD.

All subjects will be required to be off all prescription medications which could effect the PET scan, such as medications with anticholinergic effects, for two weeks to one month prior to the PET scan, and off psychotropic medication for one month.

Subjects will be cautioned not to consume alcohol, marijuana, or psychotropic drugs while on the study, nor to smoke, use caffeinated beverages, or take over-the-counter medications such as cold medications (ie: Benadryl, Sudafed) for at least 12 hours prior to the PET scan.

EXCLUSION CRITERIA:

Patients withe significant cardiovascular disease, history of alcoholism, significant head trauma, uncontrolled hypertension, diabetes, bleeding disorders or other medical conditions which would make it medically unsafe to perform any part of the PET scan or would confound data analysis.

Subjects with evidence of significant chronic disease to be accepted into the healthy control group.

Subjects must not be pregnant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1999-04; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Christie JE, Shering A, Ferguson J, Glen AI. Physostigmine and arecoline: effects of intravenous infusions in Alzheimer presenile dementia. Br J Psychiatry. 1981 Jan;138:46-50. doi: 10.1192/bjp.138.1.46. PMID 7023592
- [Background] Davis KL, Hollister LE, Overall J, Johnson A, Train K. Physostigmine: effects on cognition and affect in normal subjects. Psychopharmacology (Berl). 1976 Dec 21;51(1):23-7. doi: 10.1007/BF00426316. PMID 827772
- [Background] Davis KL, Mohs RC. Enhancement of memory processes in Alzheimer's disease with multiple-dose intravenous physostigmine. Am J Psychiatry. 1982 Nov;139(11):1421-4. doi: 10.1176/ajp.139.11.1421. PMID 6753611